CLINICAL TRIAL: NCT02148783
Title: Dopamine Receptor Imaging to Predict Response to Stimulant Therapy in Chronic TBI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment was slower than anticipated. Incomplete neuropsychological outcome measures obtained.
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ramon Diaz-Arrastia, Professor of Neurology, Uniformed Services University of the Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 402693-1; HJF grant (Other Grant/Funding Number: HJF 306136-12.01-60855)
Record Dates: First submitted 2014-05-20; First posted 2014-05-28 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury; Attention deficit and memory problems; Methylphenidate; Dopamine receptor imaging; Motivation and reward; Positron emission tomography; Transcranial magnetic stimulation
MeSH Terms: conditions — Brain Injuries, Traumatic; Attention Deficit Disorder with Hyperactivity; Memory Disorders | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- methylphenidate administration (Experimental): All participants will receive oral methylphenidate 60 mg before the second TMS study. The participants will receive oral methylphenidate 60 mg before the second PET scan. Subjects will then be treated with oral methylphenidate, using a forced titration. Dose titration will be incremental within 6 days (dose-escalation phase) , starting at 5 mg orally twice daily for 3 days, and 10 mg twice daily for the next 3 days. Then the dose will be increased to 30 mg twice daily starting from day 7 given twice daily for additional 3 weeks.
  Interventions: Drug: methylphenidate; Drug: Placebo

INTERVENTIONS:
Drug: methylphenidate — This is an open-labeled 4 week methylphenidate administration, 30 mg twice daily by mouth. Placebo and methylphenidate will also be administered as a single dose before one of the two PET and TMS sessions, in a single blinded manner (the participant will not know whether active drug or placebo was administered). PET imaging with [11C]-raclopride, a D2/D3 receptor ligand will be performed after administration of placebo or oral methylphenidate to measure endogenous DA release in TBI patients. Structural MRI will be performed before methylphenidate administration. TMS after placebo or methylphenidate will be performed to measure intracortical inhibition and dopaminergic activity.
  Other Names: Ritalin
Drug: Placebo

SUMMARY:
Deficits in memory, attention, cognitive, and executive functions are the most common disabilities after traumatic brain injury (TBI). Dopamine (DA) neurotransmission is implicated in these neural functions and dopaminergic pathways are recognized to be frequently disrupted after TBI. One of the most widely used DAergic drugs is methylphenidate (Ritalin®). Methylphenidate increases synaptic DA levels by binding to presynaptic dopamine transporters (DAT) and blocking re-uptake. PET with methylphenidate challenge to measure tonic DA release provides valuable insight into the molecular basis of attention-deficit hyperactivity disorder (ADHD) and addiction, as well as practical information regarding likely effectiveness of therapy (1). The objectives of this study are to use PET imaging with [11C]-raclopride, a D2/D3 receptor ligand, before and after administering methylphenidate, to measure endogenous DA release in patients who are experiencing problems with cognition, attention and executive function in the chronic stage after TBI. In addition, we will use TMS to test short intracortical inhibition, a gamma-aminobutyric acid receptor A (GABAA) - mediated phenomenon, which is under partial DA control, as a measure of dopaminergic activity on and off methylphenidate.

DETAILED DESCRIPTION:
* Males and females (n=30), between the ages of 18 and 55 years in the chronic stage after TBI who experience deficits in neuropsychological function from TBIs incurred 6 months after the injury, will be recruited from military treatment facilities or civilian clinics when presenting for clinical management of TBI or post-concussive symptoms.
* 1. Study participants will be evaluated using brain MRI, psychometric measures adapted from the TBI Common Data Elements, attention tests and information about details of the injury and experience of post-concussive symptoms will be recorded. Transcranial magnetic stimulation (TMS) with placebo and with methylphenidate (60 mg by mouth) challenge will be performed to predict a stimulant response.
* 2. Subjects will be studied with [11C]-raclopride PET in two imaging sessions. One session will be after administration of placebo and the other after methylphenidate, 60 mg by mouth. Both placebo and methylphenidate will be given 60 minutes prior to injection of [11C]-raclopride to allow for peak uptake of methylphenidate in the brain. The binding potential of [11C]-raclopride relative to a non-displaceable reference region (cerebellum), BPND, will be used as a measure of D2/D3 receptor availability. The difference in BPND between methylphenidate and placebo (ΔBPND) is used to measure of tonic DA release.
* 3. Subjects will then be treated with oral methylphenidate, using a forced titration up to a dose of 30 mg given twice daily for 4 weeks. At that point, the neuropsychologic tests are repeated.
* Outcome measures: The primary outcome is change in information processing speed during neuropsychologic testing.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 55 years, inclusive
* A history of having sustained a moderate or severe TBI > 6 months prior to enrollment. Evidence will be any one of the following 3 criteria:

  1. GCS 3 - 12 (GCS obtained in Emergency Room and noted in medical record)
  2. Post-traumatic amnesia > 24 hours
  3. TBI-related abnormality on neuroimaging (either CT or MRI).
* Persistent post-concussive symptoms, according to the DSM-IV Research Criteria for Post-Concussional Disorder, including:

  1. Difficulty in attention or memory.
  2. One or more of the following symptoms, which started shortly after the trauma and persist for at least three months:

     1. Fatigability
     2. Disordered sleep
     3. Changes in personality
     4. Apathy or lack of spontaneity
  3. Symptoms in criteria (a) and (b) must have their onset after trauma, or there was a significant worsening of pre-existing symptoms after trauma.
  4. Disturbance from these symptoms causes significant impairment of social or occupational functioning and represents a significant decline from previous level of functioning.
* Ability to read, write, and speak English
* Ability to give informed consent.

Exclusion Criteria:

* Evidence of penetrating brain injury.
* Contraindication to methylphenidate therapy:

  1. Known glaucoma (consistently raised intraocular pressure with or without associated optic nerve damage)
  2. Motor tics or a family history of Tourette's syndrome (diagnosed by presence of both multiple motor and one or more vocal tics over the period of a year, with no more than three consecutive tic-free months)
  3. Known hypersensitivity to methylphenidate (hives, difficulty breathing, and swelling of face, lips, tongue, or throat).
  4. Known severe anxiety or restlessness which prevents from doing day to day activities.
  5. Known preexisting hypertension, heart failure, myocardial infarction, or ventricular arrhythmia.
  6. Known preexisting psychosis, bipolar illness.
  7. History of seizures, or interictal epileptiform discharges (IEDs) on EEG in absence of seizures.
  8. Known peripheral vasculopathy, including Raynaud's phenomenon.
  9. History of drug dependence or alcoholism.
  10. Concomitant treatment with coumadin anticoagulants, anticonvulsants (e.g., phenobarbital, phenytoin, primidone), and tricyclic drugs (e.g., imipramine, clomipramine, desipramine).
  11. Concomitant therapy with monoamine oxidase inhibitors (such as Marplan (isocarboxazid), Nardil (phenelzine), Emsam (selegiline), and Parnate (tranylcypromine))
  12. Concomitant treatment with blood pressure medication (both for high and low blood pressure).
  13. Pregnancy
  14. Breastfeeding
* History or evidence of disabling pre-existing or co-existing disabling neurologic or psychiatric disorders not related to TBI, such as:

  1. Multiple sclerosis, pre- or co-existing
  2. Stroke (other than stroke at the time of TBI)
  3. Pre-existing disabling developmental disorder
  4. Pre-existing epilepsy
  5. Pre-existing major depressive disorder, aggressive behavior, hostility
  6. Pre-existing schizophrenia
* Contraindication to MRI scanning

  1. Ferromagnetic metal in the cranial cavity or eye, e.g., aneurysm clip, implanted neural stimulator, cochlear implant, or ocular foreign body
  2. Implanted cardiac pacemaker or auto-defibrillator or pump
  3. Non-removable body piercing
  4. Claustrophobia
  5. Inability to lie supine for two hours
* Contraindication to TMS, such as metal in the cranial cavity or implanted electronic hardware.
* Current participation in other interventional clinical trial
* Non-adherence to use of effective method of contraception for females of able to become pregnant for time from enrollment to the study until 2 weeks after completion of the study drug.
* Present history of alcohol and substance abuse disorder determined by DSM-IV
* Body mass index (BMI) > 30

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2014-09; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Relationship between tonic dopamine release (measured by displacement of [11C]-raclopride by oral methylphenidate) and change in processing speed between baseline and after methylphenidate treatment. | Four weeks of treatment with methylphenidate.
  Processing speed will be assessed as a composite score of the following measures:
  1. Conners Continuous Performance Test (3rd Edition)
  2. SeaShore Rhythm Test
  3. Flanker Inhibitory Control and Attention Test
  4. Pattern Comparison Processing Speed Test

SECONDARY OUTCOMES:
Relationship between D2/D3 receptor availability in ventral striatum and prefrontal cortex and neuropsychologic deficits. | Baseline visit
  Composite measure of neuropsychologic tests selected from TBI Common Data Elements.
Relationship between tonic dopamine release in the ventral striatum and prefrontal cortex with neuropsychologic deficits after TBI. | Baseline visit
  Composite measure of neuropsychologic tests selected from TBI Common Data Elements.
Relationship between D2/D3 receptor availability and functional connectivity of the prefrontal cortex with nodes of the default mode network. | Baseline visit
Relationship between TMS-induced short-interval cortical inhibition of M1 and tonic dopamine release. | Baseline visit
Test motivation and reward on and off methylphenidate in TBI patients. | Four weeks of treatment with methylphenidate.

OTHER OUTCOMES:
Explore relationship between structural connectivity (measured by Diffusion Tensor Imaging) between the ventral striatum, prefrontal cortex, and ventral tegmental area, and tonic dopamine release in patients with TBI. | Baseline visit.

CONTACTS AND LOCATIONS:
Overall Officials: Ramon R Diaz-Arrastia, MD, PhD, Study Director — Uniformed Services University / NINDS; Eric Wassermann, MD, Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health, Clinical Center., Bethesda, Maryland, United States

REFERENCES:
- [Background] Volkow ND, Wang GJ, Tomasi D, Kollins SH, Wigal TL, Newcorn JH, Telang FW, Fowler JS, Logan J, Wong CT, Swanson JM. Methylphenidate-elicited dopamine increases in ventral striatum are associated with long-term symptom improvement in adults with attention deficit hyperactivity disorder. J Neurosci. 2012 Jan 18;32(3):841-9. doi: 10.1523/JNEUROSCI.4461-11.2012. PMID 22262882
- [Background] Whyte J, Hart T, Vaccaro M, Grieb-Neff P, Risser A, Polansky M, Coslett HB. Effects of methylphenidate on attention deficits after traumatic brain injury: a multidimensional, randomized, controlled trial. Am J Phys Med Rehabil. 2004 Jun;83(6):401-20. doi: 10.1097/01.phm.0000128789.75375.d3. PMID 15166683